CLINICAL TRIAL: NCT03605251
Title: An Early Phase-II, Randomized, Double-blind, Study of TAS5315 in Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate
Brief Title: Efficacy and Safety Study of TAS5315 Compared With Placebo in Participants With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10063030
Record Dates: First submitted 2018-07-03; First posted 2018-07-30 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAS5315 low dose group (Experimental): TAS5315 low dose and Methotrexate as specified
  Interventions: Drug: TAS5315 low dose
- TAS5315 high dose group (Experimental): TAS5315 high dose and Methotrexate as specified
  Interventions: Drug: TAS5315 high dose
- Placebo group (Placebo Comparator): Placebo and Methotrexate as specified
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: TAS5315 low dose — Oral administration for 12 or 36 weeks
  Arms: TAS5315 low dose group
Drug: TAS5315 high dose — Oral administration for 12 or 36 weeks
  Arms: TAS5315 high dose group
Drug: Placebos — Oral administration for 12 weeks (At Week 12, participants in the placebo group will be assigned to TAS5315 low or high dose group)
  Arms: Placebo group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of TAS5315 in combination with methotrexate in a 12 week or 36 week in participants with rheumatoid arthritis with inadequate response to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of RA according to 2010 ACR/ EULAR rheumatoid arthritis (RA) classification criteria
* Have been treated with methotrexate (MTX) for at least 90 days prior to screening, and must be on a stable dose between 8 and 16 mg/week for at least 56 days prior to screening.
* Have an inadequate response to MTX
* Have a minimum of 6 swollen and 6 tender joints from 66/68 joint count
* Have hsCRP of ≥ 0.6 mg/dL

Exclusion Criteria:

* Have been treated with conventional synthetic disease-modifying anti-rheumatic drug, except for MTX, within 28 days prior to randomization
* Have an inadequate response to biologic disease-modifying anti-rheumatic drug or Have been treated with 2 biologic treatment
* Have been treated with Janus Kinase inhibitors or other Bruton's Tyrosine Kinase inhibitors
* Have a positive result for hepatitis B surface antigen/antibody, hepatitis B core antibody, hepatitis C virus antibody or human immunodeficiency virus antigen/antibody at screening
* Have been treated with Oral steroids at dose above 10 mg/day of prednisone or prednisone equivalents
* Have a diagnosis of Felty's syndrome
* Have a positive result of the QuantiFERON®-tuberculosis (TB) Gold test or a T-spot ®-TB test at screening
* Have a positive result of β-D-glucan at screening

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving American College of Rheumatology 20% (ACR20) response | Week 12

SECONDARY OUTCOMES:
Proportion of participants who achieve ACR20 response | Up to Week 36, except for Week 12
Proportion of participants achieving American College of Rheumatology 50% (ACR50) and American College of Rheumatology 70% (ACR70) response | Up to Week 36
Proportion of participants who achieve DAS28-hs C-ReactivePprotein (CRP) and DAS28-Erythrocyte Sedimentation Rate (ESR) for remission | Baseline, Week 12
Change from baseline in DAS28-CRP and DAS28-ESR score | Up to Week 36
Proportion of participants who achieve Clinical Disease Activity Index (CDAI) and Simplified Disease Activity Index (SDAI) for remission | Baseline, Week 12
Change from baseline in CDAI and SDAI score | Up to Week 36
Change from baseline in patient assessment score of arthritis pain | Up to Week 36
Change from baseline in patient global assessment score of arthritis | Up to Week 36
Change from baseline in physician's global assessment score of arthritis | Up to Week 36
Change from baseline in modified total sharp score | Baseline, Week 2, 4, 12
Change from baseline in Anti-cyclic Citrullinated Peptide antibody levels | Up to Week 36
Change from baseline in rheumatoid factor levels | Up to Week 36
Maximum observed plasma concentration for TAS5315 | Baseline, Week 2, 4, 12
Time to reach the maximum plasma concentration for TAS5315 | Baseline, Week 2, 4, 12
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration for TAS5315 | Baseline, Week 2, 4, 12
Incidence of adverse events and side effects as safety | Up to Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- Taiho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Takeuchi T, Tanaka S, Murata M, Tanaka Y. Irreversible covalent Bruton's tyrosine kinase inhibitor, TAS5315 versus placebo in rheumatoid arthritis patients with inadequate response to methotrexate: a randomised, double-blind, phase IIa trial. Ann Rheum Dis. 2023 Aug;82(8):1025-1034. doi: 10.1136/ard-2022-223759. Epub 2023 May 22. PMID 37217273